CLINICAL TRIAL: NCT03153839
Title: Influence of the Aquatic Physical Activity for the Neurologic Development of the Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María José Aguilar Cordero, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25/11/2016 UGR
Record Dates: First submitted 2016-12-13; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Infant Behavior; Gestational Age Over 30 Weeks
Keywords: Children; Babies; Infant; Swimming pool; Aquatic physical activity; Motor development; Neurodevelopment
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): 74 infants who will practice with their parents a programme of aquatic physical activity in a swimming pool for one year. They will be evaluated before and after the programme.
  Interventions: Behavioral: Aquatic physical activity in babies
- Control group (No Intervention): 71 infants who will not practice the programme. They only will be evaluated.

INTERVENTIONS:
Behavioral: Aquatic physical activity in babies — A programme based on four different types exercises realized in a swimming pool for twelve months.
  Before the beginning of the aquatic physical activity, the infants will be evaluated. Afther that, the study group will practise the exercises with their parents in 20 minutes sessions twice a week and when they finish the programme they will be evaluated again.
  Arms: Study group

SUMMARY:
Introduction: physical activity in infants through aquatic therapy is widely known for the later development of sensory ,cognitive and motor areas. In this way, babies will have a greater sense of freedom, pleasure and memory of the maternal uterus. In addition, the margin therapeutic safety in the water is very broad, which allows an optimal development of aquatic early stimulation programs.

Objective: To determine the relationship between aquatic physical activity in infants and the development of their psychomotor skills in their first year.

Methods: A prospective case-control study will take place for 12 months. Participating infants will be divided in two groups: an experimental group, which will be integrated by 74 babies who will participate with their parents in the aquatic physical activity programme in a heated pool (34-35ºC) and a control group with 71 babies who will not participate in the activities. The aquatic activity will consist on 20 minutes sessions twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Commitment to participate voluntarily.
* Signing informed consent to participate in the research, according to the Helsinki Declaration, updated at the 64th General Assembly, Fortaleza, Brazil, October 2013.

Exclusion Criteria:

* Babies who are born with a gestational age of less than 30 weeks.
* Baby changes that prevent physical activity.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of baby development | 12 months
  According to the Brunet-Lezine test summarized, evaluating 5 items: motor characteristics, adaptation, language, personal and social behavior and warning signs

SECONDARY OUTCOMES:
Evaluation of the development of affectivity | 12 months
  Test Q-Sort
Gestational age | 37- 42 Weeks
  Weeks of Gestation at birth
Labour alterations | 3 months
  Compiled from clinical history
Apgar at birth | 3 months
  Apgar test
Newborn data | 3 months
  Compiled from clinical history
Type of childbirth | 3 months
  Compiled from clinical history
Nutrition of the baby. | 12 months
  Lactation, formula or complementary feeding
Family demographic variables | 3 months
  Compiled from clinical history
Family history of illness. | 3 months
  Compiled from clinical history
Toxic habits of parents | 3 months
  Compiled from clinical history

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granda, Granada, Spain